CLINICAL TRIAL: NCT00563901
Title: GenHAT - Genetics of Hypertension Associated Treatments - Ancillary to ALLHAT
Brief Title: Analyzing How Genetics May Affect Response to High Blood Pressure Medications
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Texas (Other); University of Minnesota (Other)
Responsible Party: Donna K. Arnett, PhD, University of Alabama at Birmingham
Other Study IDs: 1402; R01HL063082-07A1 (NIH)
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2008-01

CONDITIONS: Hypertension; Coronary Disease; Cerebrovascular Accident
Keywords: CHD; Combined CHD; Stroke; Combined Cardiovascular Disease (CVD); Pharmacogenetics; End-Stage Renal Disease; Heart Failure; Hospitalized/Fatal Heart Failure; Angina; Coronary Revascularizations; CHD Mortality; Lisinopril; Chlorthalidone; Amlodipine; Doxazosin
MeSH Terms: conditions — Hypertension; Coronary Disease; Stroke; Kidney Failure, Chronic; Heart Failure; Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples with DNA

GROUPS / COHORTS (1):
- 1: Adults with a high risk for high blood pressure from the ALLHAT study

SUMMARY:
High blood pressure is one of the most common health problems in the United States. There are many medications to treat high blood pressure, but there is a large variance in how people respond to these medications. It is believed that genetic variations may contribute to the inconsistent treatment response. This study will use genetic analysis to determine whether particular genes interact with high blood pressure medications to modify the risk of certain cardiovascular diseases.

DETAILED DESCRIPTION:
High blood pressure affects nearly one in three individuals in the Unites States. There are many factors that can cause high blood pressure, including family history and genetic traits, kidney disease, stress, diabetes, and diet. If left untreated, high blood pressure can increase one's risk for coronary heart disease (CHD), stroke, heart attack, and heart failure. While high blood pressure can be managed with medication, people receiving medication treatment for high blood pressure are still variably at risk for CHD and other cardiovascular conditions. This risk variation may stem from varying drug reactions that are likely due to genetics. This study will use genetic analysis to determine whether particular genes interact with high blood pressure medications to modify the risk of certain cardiovascular diseases.

This is a continuation study to the antihypertensive and lipid-lowering treatment to prevent heart attack trial (ALLHAT), which included a randomized trial of the four high blood pressure drugs chlorthalidone, amlodipine, lisinopril, and doxazosin. Using samples from ALLHAT participants, this study will analyze the interactions of candidate gene pathways of relevance with medications from the ALLHAT study. Researchers will examine both single DNA building blocks and multiple genes in the candidate gene pathways and determine whether their interaction with the ALLHAT drugs modifies the risk of cardiovascular outcomes. Researchers will perform genetic analysis on 96 genetic markers using structured association testing (SAT) and false discovery rate (FDR) methods. These methods will control for population stratification and multiple testing. Finally, the study will establish a mechanism for other researchers to continue further analysis of the genetic variants examined in this study.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the ALLHAT study

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population samples will be taken from adults who are high risk for high blood pressure in the ALLHAT study, which included a randomized trial of the four high blood pressure drugs chlorthalidone, amlodipine, lisinopril, and doxazosin.
Sampling Method: Non-Probability Sample
Enrollment: 37939 (Actual)
Dates: Start 2000-09; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Candidate genes that interact with ALLHAT high blood pressure medications to modify risk of other cardiovascular conditions | Measured at completion of genetic analysis

SECONDARY OUTCOMES:
Within selected candidate genes, effect of multiple gene interactions with high blood pressure medications in modifying risk of other cardiovascular conditions | Measured at completion of genetic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Donna K. Arnett, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - University of Texas Houston, Houston, Texas

REFERENCES:
- [Background] Arnett DK, Boerwinkle E, Davis BR, Eckfeldt J, Ford CE, Black H. Pharmacogenetic approaches to hypertension therapy: design and rationale for the Genetics of Hypertension Associated Treatment (GenHAT) study. Pharmacogenomics J. 2002;2(5):309-17. doi: 10.1038/sj.tpj.6500113. PMID 12439737
- [Background] Davis BR, Ford CE, Boerwinkle E, Arnett D, Eckfeldt J, Black H. Imputing gene-treatment interactions when the genotype distribution is unknown using case-only and putative placebo analyses--a new method for the Genetics of Hypertension Associated Treatment (GenHAT) study. Stat Med. 2004 Aug 15;23(15):2413-27. doi: 10.1002/sim.1831. PMID 15273956
- [Result] Arnett DK, Davis BR, Ford CE, Boerwinkle E, Leiendecker-Foster C, Miller MB, Black H, Eckfeldt JH. Pharmacogenetic association of the angiotensin-converting enzyme insertion/deletion polymorphism on blood pressure and cardiovascular risk in relation to antihypertensive treatment: the Genetics of Hypertension-Associated Treatment (GenHAT) study. Circulation. 2005 Jun 28;111(25):3374-83. doi: 10.1161/CIRCULATIONAHA.104.504639. Epub 2005 Jun 20. PMID 15967849
- [Result] Davis BR, Arnett DK, Boerwinkle E, Ford CE, Leiendecker-Foster C, Miller MB, Black H, Eckfeldt JH. Antihypertensive therapy, the alpha-adducin polymorphism, and cardiovascular disease in high-risk hypertensive persons: the Genetics of Hypertension-Associated Treatment Study. Pharmacogenomics J. 2007 Apr;7(2):112-22. doi: 10.1038/sj.tpj.6500395. Epub 2006 May 16. PMID 16702981
- [Result] Maitland-van der Zee AH, Boerwinkle E, Arnett DK, Davis BR, Leiendecker-Foster C, Miller MB, Klungel OH, Ford CE, Eckfeldt JH. Absence of an interaction between the angiotensin-converting enzyme insertion-deletion polymorphism and pravastatin on cardiovascular disease in high-risk hypertensive patients: the Genetics of Hypertension-Associated Treatment (GenHAT) study. Am Heart J. 2007 Jan;153(1):54-8. doi: 10.1016/j.ahj.2006.10.019. PMID 17174637
- [Derived] Sherva R, Ford CE, Eckfeldt JH, Davis BR, Boerwinkle E, Arnett DK. Pharmacogenetic effect of the stromelysin (MMP3) polymorphism on stroke risk in relation to antihypertensive treatment: the genetics of hypertension associated treatment study. Stroke. 2011 Feb;42(2):330-5. doi: 10.1161/STROKEAHA.110.593798. Epub 2010 Dec 23. PMID 21183746